CLINICAL TRIAL: NCT06393335
Title: Safety and Efficacy of Metabolically Armed CD19 CAR-T Cells (Meta10-19) in the Treatment of Relapsed and/or Refractory CD19-positive B Cell Hematological Malignancies Clinical Research
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaojun Xu, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Meta10-19-005
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Acute Lymphoblastic Leukemia; Non-hodgkin Lymphoma
Keywords: Meta10-19; CAR-T Cells Therapy; CD19-positive B cell Hematological Malignancies
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Metabolically Armed CD19 CAR-T cells (Experimental): Patients undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CAR-T cells infusion. A dose of metabolically armed CD19 CAR-T cells will be infused on day 0.
  Interventions: Drug: Metabolically Armed CD19 CAR-T cells

INTERVENTIONS:
Drug: Metabolically Armed CD19 CAR-T cells — Each subject receive metabolically armed CD19 CAR- T cells by intravenous infusion.
  Other Names: Meta10-19

SUMMARY:
A Study of Metabolically Armed CD19 CAR-T Cells Therapy for Patients With Relapsed and/or Refractory CD19-positive B cell Hematological Malignancies

DETAILED DESCRIPTION:
This is a single arm, open-label study. This study is indicated for relapsed or refractory CD19-positive B cell Hematological Malignancies.

1. Main research objectives:

   To evaluate the safety and efficacy of metabolically armed CD19 CAR-T Cells in the treatment of r/r CD19-positive B cell Hematological Malignancies
2. Secondary research objectives:

   1. To evaluate the pharmacokinetic (PK) and pharmacodynamics(PD) characteristics of metabolically armed CD19 CAR-T Cells after infusion.
   2. To evaluate tumor remission after infusion of metabolically armed CD19 CAR-T Cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 6 months to 18 years old, inclusive, for both males and females.
2. The patient or their guardian voluntarily signed the informed consent.
3. Patients with relapsed or refractory CD19-positive B cell hematological malignancies:

   1. Relapsed or refractory B-ALL (meeting one of the following conditions):

      * Patients who relapse within 30 months after the initial remission, with >5% primordial cells (lymphoblast and prolymphocyte) in bone marrow morphology, confirmed by flow cytometry.
      * Patients who relapse 30 months after the initial remission and fail to achieve complete remission or show poor response to early treatment after one course of standardized induction therapy.
      * Patients who relapse after allogeneic hematopoietic stem cell transplantation (HSCT) and must undergo screening 3 months post-HSCT .
      * Patients who do not achieve CR after standardized chemotherapy, or have >1% minimal residual disease (MRD) in bone marrow after 3 months of chemotherapy.
      * Philadelphia-chromosome-positive (Ph+) patients who do not achieve CR or relapse after being treated with at least two tyrosine kinase inhibitors (TKI).
      * Patients who are not suitable candidates for allogeneic hematopoietic stem cell transplantation.
   2. Relapsed or refractory CD19+ B-NHL (meeting one of the following conditions):

      * Patients who have been treated with CD20 antibodies (such as rituximab) and at least two chemotherapy regiments, one of which should include anthracyclines.
      * After these treatments, patients experienced stable disease (SD) (with SD duration ≤12 months) or disease progression.
      * Patients who relapse after auto/allo-HSCT, or are not eligible for HSCT.
      * Patients with double-hit and triple-hit lymphoma who do not respond to second-line treatment.
4. Positive CD19 expression comfirmed by immunohistochemistry or flow cytometry.
5. For participants who had failed prior CD19-CAR T cell therapy: at least 30-days has elapsed since participant received last CD19-CAR T cell therapy.
6. Presence at least one measurable lesion at baseline, as per the initial assessment, staging and response assessment recommendations for Hodgkin's and non-Hodgkin's lymphoma (2014 edition).
7. Life expectancy ≥ 12 weeks.
8. ECOG ≤ 1.
9. Organ function:

   1. Complete blood count (CBC) test results should meet the following criteria within 24 hours before apheresis (Avoid blood/platelet transfusion, cell growth factors (except recombinant erythropoietin) and other supportive treatments within 7 days prior to the test):

      * Absolute Lymphocyte Count (ALC) ≥ 0.5×10^9 /L (except for those receiving bridging chemotherapy).
      * Platelet (PLT) ≥ 25×10^9 /L.
      * Hemoglobin (Hb) ≥ 70.0 g/L
   2. Blood biochemistry:

      * Serum creatinine (Scr) ≤ 1.5× Upper limit of normal (ULN), or Creatinine Clearance (Ccr) ≥ 40 mL/min (calculated using the Cockcroft-Gault formula).
      * Alanine aminotransferase (ALT) ≤ 2.5×ULN.
      * Aspartate aminotransferase (AST) ≤ 2.5×ULN.
      * Total bilirubin (TBIL) ≤ 2×ULN; Patients who with Gilbert-Meulengracht syndrome with TBIL ≤ 3×ULN and Direct Bilirubin (DBIL) ≤1.5×ULN may be included.
      * Amylase (AMY) and Lipase (LPS) ≤ 1.5×ULN.
      * Alkaline phosphatase (ALP) ≤ 2.5×ULN.
      * If bone or liver metastases are present, AST, ALT, ALP ≤ 5×ULN.
   3. Prothrombin time (PT) was extended ≤ 4 s, fibrinogen ≥ 1 g/L, activated partial thromboplastin time (APTT) ≤ 1.5×ULN.
   4. Pulmonary function: dyspnea ≤ CTCAE grade 1 and blood oxygen saturation (SaO2) ≥ 91% in ambient air.
10. Hemodynamic stability was determined by echocardiography or multichannel radionuclide angiography (MUGA) with a left ventricular ejection fraction (LVEF) ≥ 45％.
11. Patients taking the following medications must meet the following criteria:

    1. Steroids: Therapeutic doses of steroids must be discontinued 2 weeks prior to Meta10-19 infusion. However, physiological replacement doses of steroids are permitted, with hydrocortisone or its equivalent < 6-12mg/mm^2/day.
    2. Immunosuppressive agents: Any immunosuppressive medication must be stopped ≥ 4 weeks before signing the informed consent.
    3. Anti-proliferative therapy other than preconditioning chemotherapy should be ceased within 2 weeks prior to Meta10-19 infusion.
    4. Treatment for central nervous system (CNS) diseases must be stopped 1 week before Meta10-19 infusion (e.g., intrathecal methotrexate).
12. As determined by the researchers, patients who have recovered from the toxicity of the previous treatments, that is, the CTCAE toxicity grade is less than 1 (excluding specific toxicity of grade 2 or lower, such as hair loss, deemed irrecoverable in a short timeframe by the researchers) are suitable for receiving pretreatment chemotherapy and CAR-T cell therapy.
13. The patient should have adequate venous access for apheresis or peripheral blood collection, with no other contraindications for blood cell separation.

Exclusion Criteria:

1. Patients with a history of central nervous system (CNS) diseases other than CNS leukemia, such as seizures disorders, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
2. Patients who had received chemotherapy other than preconditioning chemotherapy within 2 weeks prior to Meta10-19 infusion.
3. Patients who have participated in other clinical trials within 30 days prior to enrollment.
4. Patients with active hepatitis B (defined as positive for hepatitis B surface antigen or hepatitis B core antibody, with concomitant hepatitis B virus DNA level > 1000 copies/ml) or hepatitis C (positive for HCV RNA).
5. Patients who are positive for HIV antibodies or treponema pallidum antibodies.
6. Patients with uncontrolled acute life-threatening bacterial, viral or fungal infections (e.g., positive blood cultures ≤ 72 hours before Meta10-19 infusion).
7. Patients with unstable angina pectoris and/or myocardial infarction within 6 months prior to enrollment..
8. Patients with history of other malignancies may be eligible for enrollment under the following conditions:

   1. Adequately treated basal or squamous cell carcinoma (requiring adequate wound healing before signing informed consent).
   2. Carcinoma in situ (DCIS) of cervical or breast cancer, which has been treated therapeutically, has shown no signs of recurrence for at least 3 years prior to the signing of the informed consent.
   3. The primary malignancy has been completely resected and in complete remission for ≥ 5 years.
9. Patients with active neuroautoimmune or inflammatory conditions (e.g., Guillian-Barre syndrome, amyotrophic lateral sclerosis).
10. Patients with other conditions deemed unsuitable for enrollment in this clinical study by the investigator.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
MTD | MTD will be determined based on DLTs observed during the first 28 days of study treatment
  Determine the Maximal Tolerable Dose(MTD)
Objective response rate (ORR) | Within 3 months following infusion of Meta10-19
  Measure Tumor response rate (including CR and PR)

SECONDARY OUTCOMES:
Concentration of CAR-T cells | Up to 12 months after CAR-T treatment
  Concentration of CAR-T cells measured by Flow cytometry after CAR-T infusion
Pharmacodynamics of CAR-T cells | Up to 28 days after infusion
  Concentration levels of CAR-T related serum cytokines such as CRP, IL-6, INF-γ at each time point

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No